CLINICAL TRIAL: NCT02469116
Title: Phase II Trial of Carboplatin Plus Docetaxel With Day 2 Pegylated G-CSF (Neulasta®) in the Front-line Treatment of Patients With Advanced Stage Ovarian Carcinoma
Brief Title: Carboplatin Plus Docetaxel With Day 2 Pegylated G-CSF (Neulasta®) in Patients With Advanced Stage Ovarian Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew financial support
Sponsor: Washington University School of Medicine (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-1023
Record Dates: First submitted 2015-06-01; First posted 2015-06-11 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Docetaxel; Carboplatin; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: (docetaxel, carboplatin, pegylated G-CSF) (Experimental): * Docetaxel intravenously over 1 hour followed by carboplatin intravenously over 30 minutes-1 hour on day 1 every 21 days for maximum of 6 cycles
  * Pegylated G-CSF on day 2 every 21 days for maximum of 6 cycles
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Pegylated G-CSF

INTERVENTIONS:
Drug: Docetaxel
  Other Names: Docefrez®; Taxotere®
Drug: Carboplatin
  Other Names: Paraplatin; CBDCA
Drug: Pegylated G-CSF
  Other Names: Neulasta®); Pegfilgrastim

SUMMARY:
In this study the investigators will be using an AUC of 6 based on creatinine clearance using the Carboplatin dosing formula used for Gynecologic Oncology Group protocols.

Given that myelosuppression was significant using the docetaxel dose of 75 mg/m*2 in the SCOTROC trial, the prophylactic use of pegylated G-CSF in this Phase II trial is warranted. The expectation would be that patients will be able to receive their cycles in a more timely fashion, with less delays, thereby allowing for improved outcomes and decreased hospitalizations due to myelosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed Stage III/IV epithelial ovarian or primary peritoneal carcinoma at time of initial diagnosis
* Treatment must start within 8 weeks of surgery
* Subjects may be measurable per RECIST criteria or evaluable for disease response by CA125. Evaluable CA 125 levels are defined as an elevated CA125 pre operatively which either remains elevated post-operatively or normalizes after surgery
* No prior chemotherapy or radiation therapy
* Age ≥ 18
* Performance Status must be ≤ 2 (ECOG)
* Peripheral neuropathy: must be ≤ grade 1
* Hematologic (minimal values)

  * Absolute neutrophil count ≥ 1,500/mm3
  * Hemoglobin ≥ 8.0 g/dl
  * Platelet count ≥ 100,000/mm3
* Hepatic

  *Total Bilirubin ≤ ULN
* AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility.

  * If alkaline phosphatase is ≤ ULN and AST or ALT is >5x ULN then the patient is not eligible
  * If alkaline phosphatase is >1x but ≤2.5 x the ULN and the AST or ALT is >1.5x the ULN then the patient is not eligible
  * If alkaline phosphatase is >2.5x but ≤5x the ULN and the AST or ALT is >1x the ULN then the patient is not eligible
  * If alkaline phosphatase is >5x the ULN then the patient is not eligible
* Renal: Creatinine (serum) less than or equal to 1.5 ULN, CTC grade 1.
* Women of childbearing potential must have a negative pregnancy test and must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

PT/PTT ≤ 1.5 x's ULN

Exclusion Criteria:

* Patients with a history of severe hypersensitivity reaction to Docetaxel or other drugs formulated with polysorbate 80.
* Women who are pregnant or breast-feeding.
* Patients who have signs of infection or who have not recovered from the effects of recent surgery
* Patients with a performance status of 3 or 4
* Patients with a second malignancy within past 5 years other than non-melanoma skin carcinoma.
* Patients who have received prior myelosuppressive chemotherapy or XRT.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-01; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Mutch, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 01/12/2006 and closed to participant enrollment on 12/01/2009.
Period: Overall Study
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade 3-4 Neutropenia as Measured by CTCAE Version 3
Time Frame: Through 30 days after completion of treatment (approximately 22 weeks)
Measure: Number; unit: participants
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Number analyzed (Participants) | 18
participants
  Grade 3 neutropenia | 4
  Grade 4 neutropenia | 0

2. Secondary Outcome: Efficacy of Regimen as Measured by CA-125 Response
Description: * Progression is defined as one of the following:
    * Patients with elevated CA-125 pretreatment and normalization of CA-125 must show evidence of CA-125 ≥ twice the upper limit of normal on two occasions at least one week apart
    * Patients with elevated CA-125 pretreatment which never normalizes must show evidence of CA-125 ≥ 2 times the nadir value OR > 50% increase from the nadir on two occasions at least one week apart,
    * Patients with CA-125 in the normal range pretreatment must show evidence of CA-125 ≥ two times the upper limit of normal on two occasions at least one week apart.
  * Complete response is defined as a CA-125 value <13 confirmed on two occasions at least 2 weeks apart.
  * Partial Response is defined as a reduction of at least 50% from the original elevated CA-125 value (original value must have been > 50), confirmed on two occasions at least 2 weeks apart.
  * Stable Disease is defined as not meeting one of the above criteria.
Time Frame: Completion of treatment (approximately 18 weeks)
Measure: Number; unit: participants
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Number analyzed (Participants) | 18
participants
  Complete response | 16
  Partial response | 1
  Stable disease | 0
  Progressive disease | 1

3. Secondary Outcome: Time to Progression (TTP)
Description: Progressive disease is at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry. Unequivocal progression of existing non-target lesions, other than pleural effusions without cytological proof of neoplastic origin, in the opinion of the treating physician within 8 weeks of study entry is also considered increasing disease (in this circumstance an explanation must be provided). In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% increase in the LD is required.
Time Frame: Completion of follow-up
Population: The sponsor withdrew funding for the study which meant there was no funding for completion of accrual, follow-up or statistical analysis.
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is the observed length of life from entry into the study to death or the date of last contact
Time Frame: Completion of follow-up
Population: as for outcome 3
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival (PFS)
Description: -Progression-Free Survival is the period from study entry until disease progression, death or date of last contact.
Time Frame: Completion of follow-up
Population: as for outcome 3
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Number analyzed (Participants) | 0

6. Secondary Outcome: Quality of Life (QoL) as Measured by FACT-O Assessment Tool
Description: * The FACT-O questionnaire consists of a Physical Well-Being Section, Social/Family Well-Being Section, Emotional Well-Being Section, Functional Well-Being Section, and Additional Concerns Section
  * Answers range from "Not at all" to "Very Much" with 0 = not at all and 4 = very much
Time Frame: Completion of follow-up
Population: as for outcome 3
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Adverse Events as Measured by Number of Events Experienced by All Participants
Time Frame: 30 days after completion of treatment (approximately 22 weeks)
Measure: Number; unit: events
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Number analyzed (Participants) | 18
events
  Low white blood cell count | 25
  Low absolute neutrophil count | 21
  Low platelet count | 47
  Low hemoglobin | 78
  Allergy/immunology | 3
  Cardiovascular | 4
  Coagulation | 1
  Constitutional symptoms | 42
  Dermatology | 64
  Endocrine | 56
  Gastrointestinal | 43
  Genitourinary/renal | 1
  Hemorrhage | 2
  Infection/febrile neutropenia | 9
  Lymphatics | 2
  Metabolic/laboratory | 74
  Musculoskeletal | 6
  Neurologic | 30
  Ocular/visual | 2
  Pain | 27
  Pulmonary | 2

ADVERSE EVENTS:
Description: Only the number of events was collected without the number of participants who experienced the event, as per standard practice in 2009. All Adverse Event data presented as an Other Pre-Specified Outcome Measure.
Arm/Group | Arm 1: (Docetaxel, Carboplatin, Pegylated G-CSF)
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes